CLINICAL TRIAL: NCT02721667
Title: Telemonitoring and Protocolized Case Management for Hypertensive Community Dwelling Seniors With Complex Care Needs
Acronym: TECHNOMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Raj Padwal, Professor, Faculty of Medicine and Dentistry, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR EH2-143571
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Hypertension
Keywords: Blood pressure; Telemonitoring; Case management; Seniors
MeSH Terms: conditions — Hypertension | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (No Intervention): Participants receive a home BP monitor, are taught how to measure home BP and are encouraged to take BP readings to appointments with their providers. In addition, they will be reminded to perform a home BP series each quarter for study outcome purposes, which will encourage self-monitoring.
  Home BP readings will be teletransmitted for data collection purposes but neither participants nor providers will have access to the these readings. High BP levels that trigger safety alerts to research personnel are the only exception - participants and their primary care providers will be made aware of these.
- Telemonitoring and Case Management (Active Comparator): Home BP series mean, trends and individual readings will be generated for use by the case manager. Participants in this arm will each be assigned a pharmacist case manager who holds full prescribing privileges and who will:
  1. Administer health behaviour modification counselling, teach BP self-monitoring, and monitor medication adherence;
  2. Review telemonitored health portal BP summaries and make medication regimen adjustments according to guideline-concordant study protocol;
  3. Fax a summary of these adjustments to the participant's primary care provider (to make them aware of treatment changes); and
  4. Facilitate communication between participants and providers.
  Interventions: Device: Telemonitoring; Other: Case Management

INTERVENTIONS:
Device: Telemonitoring — Secure, wireless transmission of home blood pressure measurements that are summarized in a secure health portal for healthcare providers use for clinical management decisions, including calculation of mean BP and graphing of temporal trends.
  Arms: Telemonitoring and Case Management
Other: Case Management — Case managers work collaboratively with patients and physicians to optimize health behaviours, monitor risk factors, implement therapeutic adjustments, encourage adherence, and coordinate follow-up care.
  Arms: Telemonitoring and Case Management

SUMMARY:
Hypertension affects over 70% of Canadians over the age of 65y. Seniors with hypertension are at high risk for cardiovascular disease and death. Most of this risk is mediated through high blood pressure (BP). However, seniors are also at risk for side effects from BP lowering medication. These can be life threatening and costly. Therefore, BP monitoring is required to ensure BP levels are in the recommended range (neither too high nor low).

Home BP monitoring can be used to ensure that BP is in the right range and is recommended for all patients with high BP. Studies in other health care systems show that, to optimally perform home monitoring, the readings should be teletransmitted (electronically sent to the care provider). Additional studies indicate that BP control improves when health care providers (usually pharmacists or nurses) are specifically assigned to review teletransmitted BP readings and, using protocols, make therapeutic adjustments. However, a study needs to be conducted within the Canadian healthcare system to prove that telemonitoring±case management is cost-effective. In addition, proof that seniors consider telemonitoring to be usable and acceptable is required.

The investigators will conduct a 200 patient randomized trial in community-dwelling seniors that will compare home BP monitoring alone to telemonitoring plus case management, to comprehensively assess cost-effectiveness, usability, and acceptability. Our partners include TeleMED, a medium sized Canadian technology company with a wealth of experience in medical data management and transmission; Pharmacare, which will provide case-management services. The study will take place in seniors' supportive living residences; by virtue of residing in these institutions, these seniors have complex care needs. This intervention, if effective, cost-effective and safe, can be widely implemented.

DETAILED DESCRIPTION:
Objective:

Assess the 'real world' effectiveness, safety and cost-effectiveness of home BP telemonitoring in combination with protocolized pharmacist case management in community-dwelling seniors with diabetes and hypertension.

Background:

Hypertension, present in over 70% of seniors, causes devastating cardiovascular complications and premature death. Despite its critical importance to health, high BP is uncontrolled in about 35% of seniors with diabetes (i.e., undertreatment). Conversely, antihypertensive drug therapy can excessively lower BP, causing serious adverse effects that warrant drug discontinuation or dose reduction (i.e., overtreatment). Both undertreatment and overtreatment lead to potentially preventable harms and thus need to be minimized.

Office BP measurements are currently used to monitor the vast majority of Canadians with hypertension; however, they are inaccurate and Canadian guidelines (May 2015) instead strongly endorse use of home BP because home readings are more accurate and more convenient to measure. Home readings can be taken in 3 ways: 1. by the patient alone (who bears responsibility for giving the readings to their provider); 2. via telemonitoring, in which readings are automatically summarized and sent to the care provider; 3. through telemonitoring plus protocolized case management, in which the summarized readings are reviewed by a case manager (usually a nurse or pharmacist) authorized to adjust treatments. Telemonitoring and case management is not being used in Canada because validation data in this country are lacking and the pre-requisite tech infrastructure does not exist. The patient alone method is being used exclusively but has many barriers and pitfalls (including failure to take the proper number of readings, report all readings, calculate mean BP, or use this information to optimally manage both inappropriately high and low BP).

Design:

In this 1-year pragmatic, prospective, randomized open label trial with blinded ascertainment of endpoints, 200 patients will be randomly assigned (1:1) to one of 2 study arms: enhanced usual care (home BP monitoring alone) or home BP telemonitoring plus protocolized case management. Randomization will be performed independent of the study team (by EPICORE Centre) through a centralized computerized concealed process, stratified by baseline BP (above versus below 140 mmHg systolic BP). Outcomes assessors and analysts will be masked to allocation status. Blinded assessment of the primary endpoint (24-hour ambulatory BP) will be performed.

Methods:

All participants will receive a validated electronic upper arm oscillometric BP device (A&D Ltd. UA-651BLE; San Jose, CA) and a set top box (a hub for wireless data transmission to a secure server). Participants without internet access will also receive a cellphone with a data plan. Pushing a single button activates the device and initiates a BP measurement, which is auto-transmitted to the set top box via a bluetooth connection. The academic research team in collaboration with TeleMED, a Canadian based telemedicine company, will build data transmission protocols (using Secure Sockets Layer [SSL] encrypted data transmission) and TeleMED will build and maintain the health portal platform.

Four BP measurements will be taken daily for 1 week (home BP series). If BP is high or low, the home BP series will be done each month until BP is in the therapeutic range. Once controlled, the protocol will be repeated every 3 months, as recommended by guidelines.

Teletransmitted BP readings will be summarized within a secure health portal using TeleMED software, which will be used to calculate an overall weekly mean. Temporal trends will be plotted. BP teletransmission will occur in all study arms but will be used differently in each.

Consecutive, consenting seniors (≥65 years) with hypertension, will be recruited from seniors supportive living residences including (but not necessarily limited to) 43 Greater Edmonton Foundation (GEF) Seniors Housing (www.gef.org) and Rosedale Seniors' Living (rosedaledevelopments.com) residences; none of these residents currently receive telemonitoring or case management. They will be followed by the study team for a period of 1 year; outcome assessments will occur at 6 and 12-months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of hypertension.
* Adequate English fluency (both verbal and written).

Exclusion Criteria:

* Systolic BP level >220 mmHg or diastolic BP level >110 mmHg on screening BP measurement (WatchBP [Microlife Corp., Widnau, Switzerland]).
* Heart failure
* Severe cognitive impairment, defined as a score of ≥ 5 on the Short Portable Mental Status Questionnaire.
* Severe depression (Patient Health Questionnaire [PHQ-8] ≥15).
* Foreshortened life expectancy (<1y).
* Participation in a concurrent cardiovascular trial.
* Currently receiving case management services for cardiovascular risk factor control.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (24-hour Ambulatory Blood Pressure Monitoring, ABPM)) | one year
  Proportion of patients with overall 24-hour ABPM in the optimal range (110-129 mmHg in patients 65-79y and 110-139 mmHg in patients 80 y or older)

SECONDARY OUTCOMES:
Blood Pressure | one year
  Change in mean 24-hour systolic and diastolic BP (overall, daytime, and nighttime), home BP and the automated BP measurements (taken at each study visit) will be examined
Postural Blood pressure changes | one year
  Change in automated BP measurements examining postural changes (sitting, supine, standing)
Antihypertensive Medications | one year
  Initiation, dosage modification and/or discontinuation of medications to control blood pressure
Incidence of Treatment-Emergent Adverse Events | one year
  Frequency of serious non-mechanical falls, syncope, hypotension, and electrolyte disturbances.
Cognition | one year
  Change in Montreal Cognitive Assessment Scale score
Cost-Effectiveness of Telemonitoring | one year
  Economic models from the health care payor perspective will be constructed and standard cost-effectiveness metrics analyzed.

OTHER OUTCOMES:
Cardiovascular Risk Factors | one year
  cholesterol, A1C, urinary albumin, smoking and other lifestyle behaviors, body mass index, waist circ
Depression | one year
  Change in Patient Health Questionnaire (PHQ-9) score
Frailty | one year
  Clinical Frailty Scale (change from baseline to one-year)
Health status | one year
  Change in EQ-5D score
Satisfaction with Medical Care | one year
  Change in Patient Satisfaction Questionnaire
Anxiety | one year
  Change in General Anxiety Disorder (GAD-2) score

CONTACTS AND LOCATIONS:
Overall Officials: Raj Padwal, MD, Msc, Principal Investigator — University of Alberta
Locations (1):
- Seniors independent living or supportive living residences in greater Edmonton., Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padwal R, McAlister FA, Wood PW, Boulanger P, Fradette M, Klarenbach S, Edwards AL, Holroyd-Leduc JM, Alagiakrishnan K, Rabi D, Majumdar SR. Telemonitoring and Protocolized Case Management for Hypertensive Community-Dwelling Seniors With Diabetes: Protocol of the TECHNOMED Randomized Controlled Trial. JMIR Res Protoc. 2016 Jun 24;5(2):e107. doi: 10.2196/resprot.5775. PMID 27343147